CLINICAL TRIAL: NCT02300181
Title: A Randomized, Double-blind, Placebo Controlled, Crossover Study to Determine the Effect of the Flour Fermentation Products by Bacillus Subtilis Var Natto DC-15 on Postprandial Glucose Profile in Prediabetic Subjects.
Brief Title: Effect of the Extract of the Flour Fermented With Bacillus Subtilis Var Natto DC-15 on Postprandial Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: NewBio Enterprise Co., ltd. (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-1051
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (flour) (Placebo Comparator): 5 placebo capsules for each test (4.88 kcal/5 cap)
  Interventions: Dietary Supplement: Placebo
- Bacillus subtilis var natto DC-15 (Experimental): 5 experimental capsules for each test (4.96 kcal/5 cap) Extract powder of the flour fermented with Bacillus subtilis var natto DC-15
  Interventions: Dietary Supplement: Bacillus subtilis var natto DC-15

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo (flour)
Dietary Supplement: Bacillus subtilis var natto DC-15
  Arms: Bacillus subtilis var natto DC-15

SUMMARY:
The purpose of the present study is to evaluate the effect of the extract of the flour fermented with Bacillus subtilis var natto DC-15 on postprandial glucose level in subjects with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose 110-125 mg/dL

Exclusion Criteria:

* Taking anti-diabetic drugs
* Taking drugs or functional food that may affect blood glucose level
* Pregnant or nursing a child
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease
* History of severe disease and/or major surgery

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Difference in plasma glucose profile including AUC and Cmax after taking 50 g carbohidrate. | Overall 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan